CLINICAL TRIAL: NCT04897750
Title: Pharmacokinetic Study of Intranasal CT001 in Children 1-17 Years of Age Undergoing Elective Surgical Procedures.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cessatech A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDC 01-0206
Record Dates: First submitted 2021-05-14; First posted 2021-05-21 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-04

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: The study population will receive a target dose of intranasal CT001 corresponding to sufentanil 0.5 mcg/kg + ketamine 0.5 mg/kg (and an additional dose 10 -15 minutes after, if needed) prior to an elective surgical, procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): a target dose of intranasal sufentanil 0,5 mcg/kg + ketamine 0,5 mg/kg, (2-4 puffs) and an additional dose if needed as premedication before placement of a PVC for induction of anaesthesia.
  Interventions: Combination Product: CT001

INTERVENTIONS:
Combination Product: CT001 — Sufentanil 0.5 mcg/kg + ketamine 0.5 mg/kg as nasal spray, followed by an additional dose 10 -15 minutes after, if needed.

SUMMARY:
This is a prospective non-randomized, open-label, single dose (and a second dose if needed), PK study in 25 children age 1-17 years. The proposed number of study participants by subset is: 8 paediatric participants 1-2 years; 8 paediatric participants >2-6 years and 9 paediatric participants >6-17 years.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric participants, age 1-17 years at the day of the surgical procedure
* Planned for elective surgical procedures (e.g. hernia, orchiopexy, gastroscopy, cystoscopy)
* ASA (American Society of Anaesthesiologists) physical status classification system score 1-2 as determined by investigator
* Planned for induction of anaesthesia by an intravenous anaesthetic agent, requiring placement of peripheral venous catheter immediately prior to the surgical procedure
* Needs premedication before induction of anaesthesia as determined by investigator
* Informed consent by the legally acceptable representative(s)
* The legally acceptable representative(s) and patients 15-17 years must be able to understand and speak local language
* A female participant who has onset of menarche is eligible to participate if she is not pregnant, not breastfeeding and agree to follow the contraceptive guidance during the treatment period for at least 7 days after administration of study treatment.

Exclusion Criteria:

* Ex-premature infant (born <37 weeks AND less than 60 weeks post conceptual age at the day of the surgical procedure)
* Mental retardation
* Abnormal nasal cavity or nasal obstruction
* Clinical contraindications to narcotic analgesia including head injury or any condition that can in the opinion of the investigator, deteriorate safety and well-being of the participants, influence PK data or optimal participation in the trial
* Medical history including substance or alcohol abuse
* Has received treatment with sufentanil and/or ketamine during the last 72 hours prior to surgery
* Has planned perioperative administration of sufentanil and/or ketamine
* Has or is suspected of having a family or personal history of malignant hyperthermia
* Has or is suspected of having allergies to ketamine or sufentanil

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Total absorption over time | 0 - 120 minutes
  Area under the concentration vs time curve
Maximum absorption | 0 - 120 minutes
  Peak concentration (Cmax)
Distribution | 120 - 240 minutes
  Volumen of distribution (Vd)
Elimination | 120 - 240 minutes
  Half life (T½)
Elimination | 120 - 240 minutes
  Clearance,

SECONDARY OUTCOMES:
Analgetic effect | 0 - 1 hour
  pain intensity by age-appropriate scale in relation to the placement of peripheral venous catheter
Sedation | 0 - 1 hour
  Assessment of sedation at the time of placement of the peripheral venous catheter using the University of Michigan Sedation Score
Feasibility, (Acceptance of intranasal administration) | 0- 4 hours
  Acceptance of the intranasal route of administration by the child, assessed by the child or legally acceptable representative or health care provider.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Classen, MD, Principal Investigator — Department of Anaesthesiology, The Juliane Marie Centre Copenhagen University Hospital
Locations (1):
- Anæstesi- og Operationsafdelingen 4013 Juliane Marie Centeret, Copenhagen, Region H, Denmark

IPD SHARING:
Plan to Share IPD: No